CLINICAL TRIAL: NCT07061418
Title: 3D Evaluation the Accuracy of Free-Handed-Countersink Guided and Fully-Guided Implant Surgery in Partially Edentulous Patients: A Clinical Trial With Quasi-experimental Study
Brief Title: 3D Evaluation of Free-handed-Countersink Guided and Fully Guided Implant Surgery in Partially Edentulous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic University of Caza, Gaza, Palestine (Other)
Responsible Party: Principal Investigator, Tayseer Afifi, Dr., Islamic University of Caza, Gaza, Palestine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC/HC/1242/23
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Partially Edentulous Jaw; Accuracy of Dental Implant Placement; Implant Deviation and Positioning Errors; Proximity to Anatomical Structures
Keywords: Countersink guided; Quasi experimental study; fully guided; Accuracy; Partially edentulous
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freehand immediate implant placement (Experimental)
  Interventions: Other: Dental Implant
- Surgery guide implant placement (Active Comparator)
  Interventions: Other: Dental Implant

INTERVENTIONS:
Other: Dental Implant — Dental implants were placed to volunteers in need of implantation in mandible, maxilla or both

SUMMARY:
This clinical trial with a quasi-experimental design investigates the accuracy of dental implant placement using three different surgical approaches: free-handed countersink guided, fully-guided, and traditional freehand techniques in partially edentulous patients. Dental implant therapy not only requires successful osseointegration but also a precise three-dimensional placement to ensure functional and esthetic outcomes. Accurate implant positioning is vital to prevent complications and ensure long-term stability. The evolution of digital technology has led to the development of computer-assisted implant surgery, enhancing surgical precision and minimizing the chances of deviation from planned positions.

In this study, implants were placed in the same patients on both sides of the jaw using two techniques for comparison - one side received a free-handed countersink guided implant, while the other used a fully-guided surgical guide. Patients included in this research were partially dentate adults with adequate oral health, bone volume, and no systemic conditions or habits that could interfere with healing. Pre-operative and post-operative cone-beam computed tomography (CBCT) scans were used to evaluate the positional accuracy of the implants.

The three-dimensional evaluation method utilized Blue Sky Plan 4 and 3D Slicer software to superimpose and analyze implant placements. Parameters such as angular deviation, crestal global deviation, apical global deviation, vertical linear deviation, lateral linear deviation, apical vertical deviation, apical lateral deviation, and distances from anatomical structures like the inferior alveolar nerve and the maxillary sinus were measured to assess placement accuracy. Measurements were taken using automatic image registration and STL superimposition of planned versus actual implant locations.

Data collected was analyzed using SPSS software. Both descriptive and inferential statistical analyses were conducted. The results aimed to determine the accuracy differences between countersink-guided and fully-guided implant techniques. The findings of this study contribute to evidence-based clinical decisions in implant dentistry by exploring if countersink-guided approaches offer comparable accuracy to fully-guided methods, thus supporting safer and more effective dental implant procedures in clinical practice.

DETAILED DESCRIPTION:
This clinical trial with a quasi-experimental study design explores the comparative accuracy of dental implant placement using three different surgical protocols in partially edentulous patients: free-handed countersink guided, fully-guided, and traditional freehand methods. The precision of implant positioning plays a pivotal role in the long-term success and aesthetics of dental implant therapy. Although osseointegration is fundamental, optimal functional and esthetic outcomes are contingent upon the precise three-dimensional positioning of the implant within the jawbone. The rationale behind this study stems from the clinical observation that improper implant placement can result in technical and biological complications, leading to treatment failure or compromised prosthetic outcomes.

The advent of digital imaging and surgical planning has revolutionized implant dentistry. Traditional radiographic stents and manual implant placement methods have been increasingly replaced by static computer-assisted implant surgery (s-CAIS), allowing for improved preoperative visualization and enhanced implant positioning accuracy. In the digital workflow, combining intraoral scans with cone-beam computed tomography (CBCT) enables clinicians to plan implant positions based on bone quality, soft tissue contours, and the spatial relationship with adjacent teeth or anatomical landmarks.

Despite these advancements, there remains a lack of clinical evidence on the performance of countersink guided protocols specifically. Countersink guided placement involves using drills designed to widen the crestal cortical bone, especially in cases of dense bone, facilitating a passive fit of the implant at the neck. This approach is typically categorized under the freehand technique but is believed to offer enhanced stability during insertion. Fully-guided surgery, in contrast, utilizes a prefabricated guide that controls each step of the drilling and implant placement process, theoretically minimizing deviation.

The study involved the recruitment of partially dentate adults who fulfilled strict inclusion criteria such as having at least six remaining teeth, good oral hygiene, sufficient bone volume for implant placement without the need for grafting, and the ability to maintain mouth opening of at least 40 mm. Patients with parafunctional habits, heavy smoking, psychiatric or systemic conditions that contraindicate implant surgery, a history of radiotherapy in the head and neck region, or younger than 18 years of age were excluded.

Each patient received two implants-one placed with the countersink guided freehand method, and the other placed using a fully-guided surgical protocol. Both procedures were performed by the same surgeon using a parallel surgical kit (Dentsply®, MIS, M4, Germany), ensuring consistency in technique and instrumentation. The implants were placed on the same day and with identical preoperative planning to eliminate inter-operator and time-related variability.

To evaluate the accuracy of implant placement, preoperative CBCT scans were taken to plan the implant location, followed by postoperative CBCT scans after implant insertion. Digital planning and analysis were conducted using Blue Sky Plan 4 software and the 3D Slicer platform. Postoperative CBCT data was processed and segmented to extract the STL file of the actual implant placement. These files were then superimposed onto the original preoperative plan using point-based automatic registration. More than twenty anatomical and reference points were marked to ensure a precise overlay, enabling a direct comparison of the actual and planned implant positions in three-dimensional space.

The primary outcome of interest was angular deviation-the angle formed between the axis of the planned implant and the axis of the inserted implant. Secondary outcomes included several linear deviations: crestal global deviation (distance between the coronal ends of the planned and placed implants), apical global deviation (distance between apical endpoints), vertical linear deviation (vertical displacement measured at the implant hexagon), lateral linear deviation (horizontal displacement along the implant axis), apical vertical deviation, and apical lateral deviation. Additionally, two anatomical safety measures were assessed: the distance from the implant to the inferior alveolar nerve in the mandible and to the maxillary sinus in the upper jaw.

These parameters were visualized and measured within the Blue Sky Plan 4 software. Measurement techniques adhered to rigorous digital protocols ensuring minimal human error and high reproducibility. The implant planned position was displayed in red, and the actual implant placement was marked in yellow, allowing for straightforward differentiation and measurement. Each deviation type was clearly outlined and labeled, enabling comprehensive analysis.

Once the measurements were collected, data entry and statistical analysis were conducted using SPSS version 22. Descriptive statistics summarized demographic and clinical characteristics of the sample. Central tendency measures provided insights into the distribution of deviation parameters. Inferential statistics included Independent t-tests for comparing mean deviation values between the countersink guided and fully-guided groups. When normality assumptions were not met, non-parametric equivalents were employed. Chi-square and Fisher's exact tests were applied for categorical variable comparisons. A 95% confidence interval was considered, with a p-value of less than 0.05 interpreted as statistically significant.

The primary objective was to determine whether the countersink guided technique demonstrated comparable accuracy to the fully-guided method. Accurate implant placement is critical not only for esthetic alignment and prosthetic function but also to prevent inadvertent injury to vital anatomical structures. Understanding whether a simpler countersink-guided approach can yield similar outcomes to more resource-intensive fully-guided surgery can have significant implications for clinical decision-making, cost-effectiveness, and treatment accessibility.

The findings of this study are expected to bridge the current knowledge gap by offering clinically derived data that supports or refutes the relative precision of countersink guided surgery. If the countersink technique proves nearly as accurate as fully-guided surgery, it may emerge as a reliable alternative in clinical scenarios where digital planning or guide fabrication is not feasible or practical. Conversely, significant deviations could reinforce the superiority of fully-guided approaches, especially in anatomically sensitive or esthetically demanding cases.

Ultimately, the goal of this research is to contribute to the evolving field of implantology by evaluating emerging surgical techniques through a robust, clinically relevant framework. This study offers valuable insights into surgical accuracy in implant dentistry and highlights the importance of precise preoperative planning, technique selection, and the integration of digital technologies to enhance patient outcomes and safety.

ELIGIBILITY:
Inclusion Criteria:

* Partially dentate adults with at least 6 remaining teeth

  * The anticipated presence of sufficient bone volume allowing for implant placement with no simultaneous bone grafting
  * Extractions within 2 months of welding.
  * Want the missing tooth to be replaced by an implant
  * Adequate related attached mucosa was found
  * Mouth opening ≥ 40 mm
  * Good oral hygiene
  * Good general health

Exclusion Criteria:

* Heavy smoking

  * Physical or psychiatric disorders preventing the implant treatment.
  * Previous radiotherapy of the head-neck region
  * Younger than 18 years

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Angular deviation | 3 months
  The primary outcome was angular deviation defined as the angle closed by the principal axis of the planned implant and the principal axis of the inserted implant in degrees.

SECONDARY OUTCOMES:
Crestal global deviation | 3 months
  **Crestal Global Deviation:** A 3D measurement of the difference between planned and actual implant positions at the bone crest. It reflects overall placement accuracy. Lower values indicate better precision.
Apical global deviation | 3 months
  **Apical Global Deviation:** A 3D measurement of the discrepancy between planned and actual implant positions at the apex. It indicates overall accuracy at the implant tip. Lower values reflect more precise placement.
Coronal Center Deviation | 3 months
  The linear distance (in millimeters) between the center of the coronal end of the planned and actual implants. It measures horizontal placement accuracy at the implant's entry point.
Apical Endpoint Deviation and Vertical Deviation | 3 months
  The apical endpoint deviation measures the distance (in mm) between the tips of the planned and inserted implants. Vertical deviation refers to the difference in height between these apical points. Both assess accuracy of depth and angular positioning.
Hexagonal Lateral Deviation | 3 months
  The lateral linear deviation is measured as the distance (in mm) between a perpendicular line on the planned implant's hexagon and a parallel line on the actual implant's hexagon. It reflects horizontal rotational or positional deviation
Apical Lateral Deviation | 3 months
  The distance (in mm) between a vertical line along the planned implant's long axis and a parallel line through the apex of the actual implant. It reflects horizontal deviation at the apical end.
Long Axis Lateral Deviation | 3 months
  The distance (in mm) between a vertical line along the long axis of the planned implant and a parallel line along the actual implant's long axis. It measures overall lateral shift of implant placement. Two anatomical parameters were also assessed alongside this measurement.
Anatomical Safety Distances (IAN and MS) | 3 months
  These measurements assess the distances (in mm) from the implant apex to the inferior alveolar nerve (IAN) in the mandible and the maxillary sinus (MS) in the maxilla. They ensure safe implant placement relative to critical anatomical structures.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Gaza, Gaza Strip, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bell CK, Sahl EF, Kim YJ, Rice DD. Accuracy of Implants Placed with Surgical Guides: Thermoplastic Versus 3D Printed. Int J Periodontics Restorative Dent. 2018 Jan/Feb;38(1):113-119. doi: 10.11607/prd.3254. PMID 29240212
- [Result] De Angelis F, Papi P, Mencio F, Rosella D, Di Carlo S, Pompa G. Implant survival and success rates in patients with risk factors: results from a long-term retrospective study with a 10 to 18 years follow-up. Eur Rev Med Pharmacol Sci. 2017 Feb;21(3):433-437. PMID 28239830
- [Result] Derks J, Hakansson J, Wennstrom JL, Tomasi C, Larsson M, Berglundh T. Effectiveness of implant therapy analyzed in a Swedish population: early and late implant loss. J Dent Res. 2015 Mar;94(3 Suppl):44S-51S. doi: 10.1177/0022034514563077. Epub 2014 Dec 11. PMID 25503901
- [Result] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT07061418/Prot_SAP_000.pdf